CLINICAL TRIAL: NCT01153802
Title: An Open Label Positron Emission Tomography Study in Healthy Male Subjects to Investigate Brain DAT and SERT Occupancy, Pharmacokinetics and Safety of Single Oral Doses ofGSK1360707, Using 11C- PE2I and 11C-DASB as PET Ligands
Brief Title: An Open Label Positron Emission Tomography Study in Healthy Male Subjects to Investigate Brain DAT and SERT Occupancy,Pharmacokinetics and Safety of Single Oral Doses of GSK1360707, Using 11C- PE2I and 11C-DASB as PET Ligands
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112773
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Depressive Disorder
Keywords: Positron Emission Tomography; serotonin; inhibitor of the neurotransmitters; safety of single oral doses; norepinephrine; dopamine
MeSH Terms: conditions — Depressive Disorder | interventions — Norepinephrine; Serotonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy Male Volunteers (Experimental): All the 12 subjects enrolled in the study were exposed to at least one dose of GSK1360707 15 mg, 30 mg, 60 mg, 90 mg, 120 mg and 150 mg. All the subjects completed the study. The initial dose, given in the study as a single-dose was 15 mg GSK1360707. The remaining subjects were dosed either as a single or split dose, as determined by the PET and tolerability data collected in the preceding subjects. The total dose did not exceed 150 mg per day, the maximum total dose given in the FTIH study.
  Interventions: Drug: GSK1360707 is a potent re-uptake inhibitor of the neurotransmitters dopamine, norepinephrine and serotonin

INTERVENTIONS:
Drug: GSK1360707 is a potent re-uptake inhibitor of the neurotransmitters dopamine, norepinephrine and serotonin — This is an open label, adaptive design, daily dosing, non-randomized PET occupancy study in healthy adult males.A range of doses may be evaluated. The initial dose, given in the study as a single dose was 150mg GSK1360707. The remaining subjects will be dosed either as a single or split dose, as determined by the PET and tolerability data collected in the preceding subjects. The total dose will not exceed 150mg per day, the maximum total dose given in the FTIH study.If dosing is conducted as a single dose, the dose will be administered after the baseline scan, If a dosing is performed in a split dose manner, dosing will occur after the baseline scan, and up to 12 hours later. The time period between doses will be determined by emerging PET occupancy data.
  Subsequent doses, if any, will be chosen based on the observed scan results. No single dose, or total dose split over 2 dosing sessions, will exceed the maximum dose in the FTIH study.

SUMMARY:
GSK1360707 is a potent re-uptake inhibitor of the neurotransmitters dopamine, norepinephrine and serotonin. This is a single dose PET study in healthy subjects.A final analyses of safety data following exposure to single oral doses, from the first time in human study, with GSK1360707 has demonstrated that the compound is well tolerated up to a dose of 150mg. This imaging study will be an open label, non-randomised PET occupancy study using healthy male volunteers. The degree and time course of DAT and SERT occupancy by GSK1360707 will be determined. The PK/PD relationship between plasma concentrations of GSK1360707 and DAT and SERT occupancy will be described.This protocol amendment includes the flexibility to split the total dose into two doses e.g. 120mg per day could be split into two doses of 60mg. Splitting the total dose is most likely required to maintain therapeutic occupancy on the transporters over the course of the day; in addition it is expected that splitting the dose may reduce effects on vital signs. Therefore collecting data following split dosing will enable best predictions of therapeutic doses to be progressed in subsequent clinical studies.

DETAILED DESCRIPTION:
GSK1360707 has been shown to exhibit pharmacological action in a wide array of in vivo models for dopaminergic activity and has been shown to significantly increase levels of the three neurotransmitters in the frontal cortex and nucleus accumbens in rats.

GSK1360707 has demonstrated antidepressant-like effects in the forced swimming test after oral administration in mice and rats. Inhibition of the three monoamines, alone or in some combination, has been implicated in the mechanism of action for currently marketed antidepressants (e.g., paroxetine [selective serotonin reuptake inhibitor], venlafaxine [serotonin and norepinephrine reuptake inhibitor], and bupropion [selective dopamine and norepinephrine reuptake inhibitor]). The known effectiveness of compounds that enhance dopaminergic, serotonergic, and/or norepinephrine activity in the treatment of depression, combined with the pre-clinical data for GSK1360707, suggests that GSK1360707 may be an effective treatment for Major Depressive Disorder (MDD). GSK1360707 has recently completed a FTIH single dose, dose escalation study in healthy young subjects (study SNV111914). The highest single dose studied was 150 mg. Single doses up to and including 150 mg were generally well-tolerated. In the FTIH study, apparent dose-dependent increases in diastolic and systolic blood pressure were observed in the dose range of 60 - 150 mg. The maximum increase in blood pressure occurred at approximately Tmax and generally continued for less than 6 h from Tmax. Preliminary data indicated, for systolic blood pressure, the maximum mean value postdose was 135 mmHg (150mg, 6 h post-dose), the maximum individual value was 164 mmHg (60mg, 3 h post-dose). For diastolic blood pressure the maximum mean value post-dose was 79 mmHg (150mg) and the maximum individual value was 113 mmHg (30mg dose). The levels of blood pressure attained post-dose with GSK1360707 is similar to the levels which occur in middle-aged men and women who were healthy or had stable cardiovascular conditions during sexual activity and exercise on treadmill [Palmeri, 2007]. This study constitutes the second clinical investigation of this compound, and will be a PET investigation of a total dose of GSK1360707 in healthy male subjects; this study will also include assessment of the pharmacokinetic parameters of GSK1360707 as well as an assessment of safety and tolerability. For serotonin reuptake inhibitors (as a class) therapeutic effects are achieved after chronic treatment generally when SERT occupancy is ≥ 80% [Meyer, 2004], therapeutic effects mediated by DAT inhibition are generally achieved when occupancy is in the region of 30% [Volkow, 2005], and abuse liability is usually avoided when DAT inhibition is <50% and there is an appropriately slow brain kinetic [Volkow, 2005]. As in vitro affinity data is not always consistent with in vivo data, information derived from in vivo assessments of target occupancy have the potential to greatly enhance the process of dose selection for phase IIa, and prediction of abuse liability. With that in mind a PET study has been conducted in Papio Anubis using [11C] DASB (a SERT ligand) and [11C]PE2I (a DAT ligand) to determine the relative in vivo affinities of GSK1360707 at SERT and DAT, and the time course of occupancy of GSK1360707 at SERT and DAT. In Papio Anubis GSK1360707 blocked both the [11C] DASB and [11C] PE2I signals indicating brain penetrancy and target binding in vivo. The in vivo affinities of GSK1360707 for DAT and SERT were found to be equivalent (EC50 ~ = 20 ng/ml @ 15 min post dose; EC50 ~ = 10 ng/ml @ 2-2.5 hr post dose), and as was the time course of GSK1360707 washout inferred from the occupancy data (t1/2 of effective free concentration = 3 hr). The lack of a suitable PET radioligand means that the degree of NAT [NET] occupancy exhibited by GSK1360707 cannot be assessed in this study. This human study will use an adaptive design to assess the time course of plasma exposure-DAT and SERT occupancy relationship in humans. The data will be used to aid dose selection for future studies. The prediction of the effective exposure in man was based on transporter occupancy [also referred to in some places as RO or receptor occupancy] (RO) due to the poor predictive power of the animal disease model (forced swimming test in rat).Predictions of human therapeutic dose for GSK1360707 are based on dissociation constant (pKi) for human SERT and DAT transporters, on transporter occupancies of GSK1360707 observed in preclinical PET studies, and on experience with our lead TRUI, GSK372475. Exposure to GSK1360707 is linear with dose and the compound shows a Tmax of approximately 2 hours, and a Cmax of approximately 50ng/mL at the highest tolerated dose of 150mg; a short terminal half-life was calculated (in the range 5-6 hours) so that plasma concentrations at 24 hours were close to the lower limit of detection (1ng/mL) or not quantifiable at all doses tested.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the
* Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.

  2.Systolic blood pressure <140 mmHg, diastolic blood pressure <90 mmHg and heart rate <90 beats/min.

  3. Male subjects between 35-55 years of age. 4.Male subjects must agree to use one of the contraception methods as listed in Section 8.1.

  5.Body Mass Index (BMI) within the range 19 - 30 kg/m2 (inclusive) at screening visit.

  6. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form 7.QTcB or QTcF < 450 msec (if the first QTcB reading exceeds the limits above, perform two more ECGs separated at least 5 min apart. Then take the average of the three QTcB to determine if the average satisfies the above criteria).

Exclusion Criteria:

* 1.Evidence or history of clinically significant hematological, renal, urinary / prostatic, endocrine, pulmonary, gastrointestinal, cardiovascular or other heart disease, glaucoma, diabetes, hepatic, neurologic (e.g. including but not limited to seizures, stroke, cerebrovascular disease or other brain conditions), or allergic disease (except for untreated, asymptomatic, seasonal allergies at time of dosing).

  2. Psychiatric illness currently or within the past year, or any lifetime history of bipolar disorder, major depressive disorder, anxiety disorder, schizophrenia or other psychotic disorder, or substance abuse or dependence (except past history of nicotine abuse/dependence if >6 months prior to screening.

  3. Subjects who, in the investigator's judgment, pose a suicidal or homicidal risk, or any subject with a history of suicidal or homicidal attempts or behaviour.

  4. The subject has a positive pre-study drug/alcohol screen. 5. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.

  6. A positive test for HIV antibody. 7. History of regular excessive alcohol consumption within 6 months of the study defined as: an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units. One unit is equivalent to a half-pint (220mL) of beer or 1 (25mL) measure of spirits or 1 glass (125mL) of wine. 8. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days , 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).

  9. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

  10. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.

  11. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor contraindicates their participation. 12. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.

  13. Unwillingness or inability to follow the procedures outlined in the protocol.

  14. Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.

  15. Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication. 16. Controlled or uncontrolled hypertension, or systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥ 90 mmHg at screening or prior to the first dose of study medication.

  17. Previous inclusion in a research and/or medical protocol involving nuclear medicine, PET or radiological investigations with significant radiation burden (a significant radiation burden being defined as ICRP category IIb or above: No more than 10 mSv in addition to natural background radiation, in the previous 3 years including the dose from this study).

  18. History of, or suffers from, claustrophobia or feels that he will be unable to lie still on his back in the PET or MRI scanner for a period of 1-2 hours.

  19. Presence of a cardiac pacemaker or other electronic device or ferromagnetic metal foreign bodies as assessed by a standard pre-MRI questionnaire.

  20. Subjects who are smokers will be excluded from this study.

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-04-03 (Actual); Primary Completion 2009-10-12 (Actual); Study Completion 2009-10-12 (Actual)

PRIMARY OUTCOMES:
To estimate the degree of DAT occupancy in brain regions of interest (ROIs)following oral doses of GSK1360707 in healthy male subjects-To estimate the degree of SERT occupancy in brain ROIs following total oral doses of GSK1360707 in healthy male subject | 6-7 weeks.
To evaluate the relationship between the plasma concentration and the resultant DAT occupancy by GSK1360707.To evaluate the relationship between the plasma concentration and the resultant SERT occupancy by GSK1360707. | 6 - 7 weeks

SECONDARY OUTCOMES:
To further assess the safety and tolerability of total oral doses of GSK1360707 including the maximal tolerated dose in the FTIH study (150 mg PO)-To further assess the pharmacokinetics of GSK1360707 in healthy male subjects | 6-7 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Comley RA, Salinas CA, Slifstein M, Petrone M, Marzano C, Bennacef I, Shotbolt P, Van der Aart J, Neve M, Iavarone L, Gomeni R, Laruelle M, Gray FA, Gunn RN, Rabiner EA. Monoamine transporter occupancy of a novel triple reuptake inhibitor in baboons and humans using positron emission tomography. J Pharmacol Exp Ther. 2013 Aug;346(2):311-7. doi: 10.1124/jpet.112.202895. Epub 2013 May 17. PMID 23685546
- See also: Results for study 112773 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/112773?search=study&search_terms=112773#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 112773 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112773 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112773 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112773 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112773 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112773 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112773 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register